CLINICAL TRIAL: NCT00574925
Title: Randomized, Double-Blind, Placebo-Controlled Multicenter Study to Assess Management Strategies for the Use of Esomeprazole (Nexium) in Helicobacter Pylori Infected Patients With Gastroesophageal Reflux Disease (GERD)
Brief Title: Study to Assess Management Strategies for the Use of Esomeprazole (Nexium) in Helicobacter Pylori Infected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACH-QBE-0201
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Last update posted 2007-12-18 (Estimated); Status verified 2007-12

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: H. pylori
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Esomeprazole

SUMMARY:
The primary objective of this study is to investigate whether eradication treatment of Helicobacter pylori followed by therapy with esomeprazole for a total of 8 weeks extends the time to relapse in patients with gastroesophageal reflux disease (GERD).

A relapse is defined by two consecutive symptom scores of the Eraflux questionnaire within 14 days that are equal or above the critical value of 25.

The secondary objectives are

1. To compare the time to relapse in the two H. pylori positive study groups with the H. pylori negative control group
2. To compare the pattern of inflammation and atrophy in the two H. pylori positive treatment groups with the naturally H. pylori negative control group at relapse.
3. All the above objectives analyzed for the efficacy subset that is the per-protocol patients broken down by effective H. pylori-eradication.

Secondary endpoints will be analyzed by the following parameters and their interactions:

1. Treatment : Eradicated, Non-eradicated, Hp-negative control
2. Esophagitis at study start: grades 0, A/B and C/D
3. Gender
4. Alcohol intake
5. NSAID/ASA intake (for histological results)

   * Trial with medicinal product

ELIGIBILITY:
Inclusion criteria:

For inclusion in the study the subject must fulfill all of the following criteria:

1. Patients aged between 18 and 70 years.
2. Chronic symptoms (>8 weeks) suggestive for GERD, as defined in Table 2 with or without reflux esophagitis grade A-D (Los Angeles classification)
3. Indication for endoscopy due to GERD symptoms is given
4. Written informed consent

Table 2: Lead GERD criteria

For inclusion in the study, all of the following lead GERD criteria should hold:

* At least one of the symptoms heartburn or regurgitation.
* At least 8 weeks ongoing symptoms.
* At least 3 times a week.
* At least moderate intensity, corresponding to light impairment in daily life and occasional need for drugs.

Exclusion criteria:

Any of the following is regarded as a criterion for exclusion from the study:

1. Severe organic esophageal disease other than reflux esophagitis (e.g. carcinoma, esophageal stenosis).
2. Gastric or duodenal ulcers
3. Patients with visible Barrett's mucosa; no histological confirmation is required for exclusion
4. History of previous esophageal or gastric surgery
5. Alcohol or drug abuse
6. Severe organic or psychiatric disease
7. Pregnancy or lactation
8. Women with child-bearing potential if no medically accepted contraceptive measures are used
9. Contra-indication to amoxicillin, clarithromycin or esomeprazole (Nexium)
10. Need for concomitant medication which could interfere with the investigational products (substrates of CYP3A4)
11. Suspected or confirmed poor compliance
12. Participation in a clinical study within 8 weeks prior to enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2003-11; Study Completion 2007-10

CONTACTS AND LOCATIONS:
Overall Officials: Werner Schwizer, MD, Principal Investigator — UniversitaetsSpital Zuerich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Schwizer W, Menne D, Schutze K, Vieth M, Goergens R, Malfertheiner P, Leodolter A, Fried M, Fox MR. The effect of Helicobacter pylori infection and eradication in patients with gastro-oesophageal reflux disease: A parallel-group, double-blind, placebo-controlled multicentre study. United European Gastroenterol J. 2013 Aug;1(4):226-35. doi: 10.1177/2050640613484020. PMID 24917966